CLINICAL TRIAL: NCT04031794
Title: Extracorporeal Membrane Oxygenator (ECMO) for Critically Ill Patients With Respiratory Failure and/or Circulatory Failure
Brief Title: ECMO for Critically Ill Patients With Respiratory Failure and/or Circulatory Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: Si 203/2018
Record Dates: First submitted 2019-07-22; First posted 2019-07-24 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Severe Acute Respiratory Distress Syndrome; Refractory Hypoxemia
Keywords: Veno-venous ECMO; Severe ARDS; Refractory Hypoxemia
MeSH Terms: conditions — Respiratory Distress Syndrome; Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conventional ARDS treatment group: Patients who they or their 1st degree relative refuse to initiate ECMO. They will receive conventional ARDS treatment.
- ECMO group: Patients who ECMO is initiated for treat refractory hypoxemia. They will receive conventional ARDS treatment and ECMO support
  Interventions: Device: Extra Corporeal Membrane Oxygenator (ECMO)

INTERVENTIONS:
Device: Extra Corporeal Membrane Oxygenator (ECMO) — Two cannular will be inserted via femoral vein or internal jugular vein and connect with blood pump and membrane oxygenation.
  Groups: ECMO group

SUMMARY:
Extracorporeal membrane oxygenation (ECMO) had been used to treat refractory hypoxemia associated with acute respiratory distress syndrome (ARDS). There were reported good outcome associated with ECMO for ARDS caused by influenza infection from several ECMO centers. However, the outcome of ECMO support in lower ECMO experience center had not been evaluated. This study aimed to evaluate the outcome of ECMO, comparing with conventional treatment among severe hypoxemic ARDS patients who were admitted in limited ECMO experience hospital.

DETAILED DESCRIPTION:
This registry enroll refractory hypoxemia ARDS patients who met the criteria for veno-venous ECMO, according to 2013 Extracorporeal Life Support Organization (ELSO) guideline criteria. The definition of refractory hypoxemia was partial pressure of oxygen:fraction of inspire oxygen (PaO2/FiO2) <100 with fraction of inspire oxygen (FiO2) >90% despite optimal mechanical ventilator support for at least 2 hours.

The ECMO team was alerted for patient evaluation. The patients, who did not consider as ECMO candidate, due to their underlying condition of terminally illness, were excluded.

The decision to initiate ECMO, or not, is dependent on the conference included the patient or the patient first relative, the attending physician and the ECMO team physicians.

Patients who ECMO is initiated will be classified into ECMO group. Patients who they or their 1st degree relative do not agree for ECMO initiation will be treated according to standard treatment for ARDS, and classified in non-ECMO group.

The patients in both groups will be follow up until they are discharged from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed ARDS according to Berlin criteria
* Refractory hypoxemia: PaO2/FiO2 <100 with FiO2 >90% despite optimal mechanical ventilator support and paralytic agent infusion
* Hypoxemia persist for at least 2 hours

Exclusion Criteria:

* Terminally ill patient
* Patient who sign for do not resuscitation
* Metastatic malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult severe ARDS with refractory hypoxemia
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-07-22 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Hospital outcome | at least 90 days
  Patient survive until discharge

SECONDARY OUTCOMES:
28 days mortality | 28 days
  Patient who dead before 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Surat Tongyoo, Dr., Principal Investigator — Mahidol University
Locations (1):
- Siriraj Hospital, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with no patient identified number.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available per request
Access Criteria: For meta-analysis

REFERENCES:
- [Background] Australia and New Zealand Extracorporeal Membrane Oxygenation (ANZ ECMO) Influenza Investigators; Davies A, Jones D, Bailey M, Beca J, Bellomo R, Blackwell N, Forrest P, Gattas D, Granger E, Herkes R, Jackson A, McGuinness S, Nair P, Pellegrino V, Pettila V, Plunkett B, Pye R, Torzillo P, Webb S, Wilson M, Ziegenfuss M. Extracorporeal Membrane Oxygenation for 2009 Influenza A(H1N1) Acute Respiratory Distress Syndrome. JAMA. 2009 Nov 4;302(17):1888-95. doi: 10.1001/jama.2009.1535. Epub 2009 Oct 12. PMID 19822628
- [Background] Noah MA, Peek GJ, Finney SJ, Griffiths MJ, Harrison DA, Grieve R, Sadique MZ, Sekhon JS, McAuley DF, Firmin RK, Harvey C, Cordingley JJ, Price S, Vuylsteke A, Jenkins DP, Noble DW, Bloomfield R, Walsh TS, Perkins GD, Menon D, Taylor BL, Rowan KM. Referral to an extracorporeal membrane oxygenation center and mortality among patients with severe 2009 influenza A(H1N1). JAMA. 2011 Oct 19;306(15):1659-68. doi: 10.1001/jama.2011.1471. Epub 2011 Oct 5. PMID 21976615
- [Background] Peek GJ, Mugford M, Tiruvoipati R, Wilson A, Allen E, Thalanany MM, Hibbert CL, Truesdale A, Clemens F, Cooper N, Firmin RK, Elbourne D; CESAR trial collaboration. Efficacy and economic assessment of conventional ventilatory support versus extracorporeal membrane oxygenation for severe adult respiratory failure (CESAR): a multicentre randomised controlled trial. Lancet. 2009 Oct 17;374(9698):1351-63. doi: 10.1016/S0140-6736(09)61069-2. Epub 2009 Sep 15. PMID 19762075
- [Derived] Tongyoo S, Chanthawatthanarak S, Permpikul C, Ratanarat R, Promsin P, Kongsayreepong S. Extracorporeal membrane oxygenation (ECMO) support for acute hypoxemic respiratory failure patients: outcomes and predictive factors. J Thorac Dis. 2022 Feb;14(2):371-380. doi: 10.21037/jtd-21-1460. PMID 35280476
- [Derived] Tongyoo S, Permpikul C, Sucher S, Thomrongpairoj P, Poompichet A, Ratanarat R, Chierakul N. Venovenous extracorporeal membrane oxygenation versus conventional mechanical ventilation to treat refractory hypoxemia in patients with acute respiratory distress syndrome: a retrospective cohort study. J Int Med Res. 2020 Jun;48(6):300060520935704. doi: 10.1177/0300060520935704. PMID 32603248